CLINICAL TRIAL: NCT00975585
Title: Clinical Evaluation of Two Silicone Hydrogel Frequent Replacement Contact Lenses
Brief Title: Clinical Performance Comparison of Two Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0907; PHNX-518
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2011-03-22 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A both eyes (Active Comparator): soft contact lens worn daily for 2 weeks, with a 2-week replacement regimen.
  Interventions: Device: senofilcon A
- lotrafilcon B both eyes (Active Comparator): soft contact lens worn daily for 4 weeks, with a 4-week replacement regimen
  Interventions: Device: lotrafilcon B

INTERVENTIONS:
Device: senofilcon A — soft contact lens, 2-week replacement indicated
  Arms: senofilcon A both eyes
Device: lotrafilcon B — soft contact lens with a 4-week replacement indicated.
  Arms: lotrafilcon B both eyes

SUMMARY:
The purpose of this study is to compare the clinical performance of two contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Existing daily soft lens wearer.
* Require a distance visual correction in both eyes.
* Have a contact lens spherical distance refraction between -1.00D and -6.00D.
* Have refractive astigmatism less than or equal to 1.00D in both eyes.
* Achieve 20/30 or better corrected distance acuity.
* Have normal eyes with no evidence of abnormality or disease.

Exclusion Criteria:

* Requires presbyopic correction.
* Requires ocular medications.
* Grade 3 or 4 ocular abnormalities.
* Grade 3 corneal staining in more than one region.
* Has had refractive surgery.
* Any other injury or ocular surgery within 8 weeks prior to study enrollment.
* Has abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Has keratoconus or other corneal irregularity.
* Polymethyl methacrylate (PMMA), Hybrid or Rigid Gas Permeable (RGP) wear in the previous 8 weeks.
* Wears habitual contact lenses that are toric, multifocal or worn extended wear.
* Any systemic illness which would contraindicate lens wear or the medical treatment of would affect vision or successful lens wear.
* Diabetic.
* Infectious or immunosuppressive disease.
* History of chronic eye disease (e.g glaucoma or age related macular degeneration).
* Pregnancy, lactation or planning pregnancy at time of enrollment.
* Participation in any concurrent clinical trial or in another trial in the last 30 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 379 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2009-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila, B Hickson-Curran, BSc, MCOptom, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (24):
- United States (24):
  - North Little Rock, Arkansas
  - Campbell, California
  - Colorado Springs, Colorado
  - Jacksonville, Florida
  - Miami, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Blue Springs, Missouri
  - New York, New York
  - Chagrin Falls, Ohio
  - North Olmsted, Ohio
  - Warren, Ohio
  - State College, Pennsylvania
  - Warwick, Rhode Island
  - Chamberlain, South Dakota
  - Hot Springs, South Dakota
  - Bartlett, Tennessee
  - Brentwood, Tennessee
  - Memphis, Tennessee
  - Tyler, Texas
  - Burlington, Vermont
  - West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A; Lotrafilcon B: contact lens
Period: Overall Study
Arm/Group | Senofilcon A | Lotrafilcon B
Started | 184 | 195
Completed | 177 | 183
Not Completed | 7 | 12
Not completed — Adverse Event | 0 | 4
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lens issue | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A | Lotrafilcon B | Total
Number analyzed (Participants) | 184 | 195 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (7.0) | 29.3 (6.9) | 29.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 136 | 261
  Male | 59 | 59 | 118
Region of Enrollment [Number; unit: participants]
  United States | 184 | 195 | 379

OUTCOME MEASURES:

1. Primary Outcome: Average Corneal Staining
Description: The overall score is the average of the total scores of each of five regions of the cornea. The minimum average score is 0 and the maximum average score is 3. Corneal surface abnormality as indicated by the severity of staining over five regions of the cornea (central, superior, inferior, nasal and temporal) was assessed by the investigator using the following scale: 0=none, 1=slight, 2=moderate, 3=severe.
Time Frame: 2 weeks
Population: Analysis included all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 177 | 183
units on a scale | 0.157 (0.018) | 0.170 (0.018)
Statistical Analysis 1: Comparison: Senofilcon A vs Lotrafilcon B; The alternative hypothesis is that senofilcon A contact lenses have non-inferior (less than or equal to) average corneal staining than lotrafilcon B after two weeks of wear; Test type: Non-Inferiority or Equivalence — Margin = 0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.014, 97.46% CI 2-sided [-0.058 to 0.031], Standard Error of Mean 0.020 — The mean difference is calculated as senofilcon A minus lotrafilcon B. Analysis is adjusted for lens type, site, lens type by site interaction as fixed effects, subject and eye nested within subject as random effects

2. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by the investigator using the Snellen chart and converted to the logarithm of the minimum angle of resolution (logMAR). logMAR ideal is 0.0 and represents 20/20 Snellen visual acuity. logMAR values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: logMAR units
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 177 | 183
logMAR units | -0.012 (0.003) | -0.002 (0.003)
Statistical Analysis 1: Comparison: Senofilcon A vs Lotrafilcon B; The alternative hypothesis is that senofilcon A contact lenses are non-inferior (less than or equal to)in visual acuity to lotrafilcon B contact lenses after two weeks of wear; Test type: Non-Inferiority or Equivalence — Margin = 0.25; Mixed Models Analysis; Mean Difference (Final Values) = -0.010, 97.46% CI 2-sided [-0.021 to -0.010], Standard Error of Mean 0.005 — The mean difference is calculated as senofilcon A minus lotrafilcon B. Analysis adjusted for lens type, site, lens type by site interaction as fixed effects, subject and eye nested within subject as random effects

3. Primary Outcome: Overall Comfort
Description: After two weeks of wear, subjects responded to a phone survey question regarding overall comfort of the study contact lenses (senofilcon A and lotrafilcon B) using the following scale: 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: 2 weeks
Population: Analysis includes subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 177 | 183
units on a scale | 3.938 (0.090) | 3.536 (0.091)
Statistical Analysis 1: Comparison: Senofilcon A vs Lotrafilcon B; The alternative hypothesis is that senofilcon A contact lenses have a higher rating of overall comfort than lotrafilcon B after two weeks of wear; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.402, 97.46% CI 2-sided [0.117 to 0.402], Standard Error of Mean 0.127 — The mean difference is calculated as senofilcon A minus lotrafilcon B. Analysis adjusted for lens type, site, lens type by site interaction as fixed effects, subject as random effects

4. Primary Outcome: Overall Comfort
Description: After four weeks of wear, subjects responded to a phone survey question regarding overall comfort of the study contact lenses (lotrafilcon B)using the following scale: 5=excellent, 4=very good, 3=good, 2=fair, 1=poor.
Time Frame: 2 weeks and 4 weeks
Population: Analysis includes all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Lotrafilcon B at 2 Weeks: lotrafilcon B contact lens after two weeks of wear
- Lotrafilcon B at 4 Weeks: lotrafilcon B contact lens after four weeks of wear
Arm/Group | Lotrafilcon B at 2 Weeks | Lotrafilcon B at 4 Weeks
Number analyzed (Participants) | 183 | 183
units on a scale | 3.534 (0.111) | 3.436 (0.118)
Statistical Analysis 1: Comparison: Lotrafilcon B at 2 Weeks vs Lotrafilcon B at 4 Weeks; The alternative hypothesis is that lotrafilcon B contact lenses have a lower rating of overall comfort after 4 weeks of wear compared to after 2 weeks of wear; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.098, 97.46% CI 2-sided [-0.218 to 0.098], Standard Error of Mean 0.141 — The mean difference is lotrafilcon B at 2 weeks minus lotrafilcon B at 4 weeks. Analysis adjusted for duration of wear, stie, duration of wear by site interaction as fixed effects, subject as random effects

5. Secondary Outcome: Limbal Redness
Description: The investigator assessed limbal redness using the following scale: 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: 2 weeks
Population: Analysis includes subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 177 | 183
units on a scale | 0.376 (0.031) | 0.499 (0.030)
Statistical Analysis 1: Comparison: Senofilcon A vs Lotrafilcon B; The alternative hypothesis is that senofilcon A contact lenses are non-inferior in limbal redness 5 to lotrafilcon B contact lenses after two weeks of wear; Test type: Non-Inferiority or Equivalence — Margin = 0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.123, 98.2% CI 2-sided [-0.123 to -0.051], Standard Error of Mean 0.030 — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Bulbar Redness
Description: The investigator assessed bulbar redness using the following scale: 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe
Time Frame: 2 weeks
Population: Analysis includes subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 177 | 183
units on a scale | 0.465 (0.031) | 0.532 (0.030)
Statistical Analysis 1: Comparison: Senofilcon A vs Lotrafilcon B; The alternative hypothesis is that senofilcon A contact lenses are non-inferior in bulbar redness to lotrafilcon B contact lenses after two weeks of wear; Test type: Non-Inferiority or Equivalence — Margin = 0.5; Mixed Models Analysis; Mean Difference (Final Values) = -0.068, 98.2% CI 2-sided [-0.068 to 0.008], Standard Error of Mean 0.032 — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Symptoms of Dryness
Description: Subjects responded to a phone survey question regarding the frequency of the sensation of dryness while wearing the study contact lenses using the following scale: 1=Extreme, 2=Moderate, 3=Slight, 4=None
Time Frame: 2 weeks
Population: Analysis includes subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 177 | 183
units on a scale | 2.003 (0.087) | 2.414 (0.088)
Statistical Analysis 1: Comparison: Senofilcon A vs Lotrafilcon B; The alternative hypothesis is that senofilcon A contact lenses have less frequency of dryness than lotrafilcon B contact lenes after two weeks of wear; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.411, 98.2% CI 2-sided [-0.411 to -0.117], Standard Error of Mean 0.124 — The mean difference is calculated as senofilcon A minus lotrafilcon B. Analysis adjusted for lens type, site, lens type by stie interaction as fixed effects, subject as random effects

ADVERSE EVENTS:
Arm/Group | Senofilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/195
Other Adverse Events (participants affected / at risk) | 0/184 | 0/195

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the PI will provide SPONSOR with at least sixty (60) days for review of a manuscript. Notwithstanding the foregoing, no paper that incorporates SPONSOR Confidential Information will be submitted for publication without SPONSOR's prior written consent. If requested in writing, the PI will withhold such publication for up to an additional sixty (60) days to allow for filing of a patent application.